CLINICAL TRIAL: NCT05038696
Title: Chimeric-Antigen Receptor (CAR) T-Cell Therapy Using Multiple CARs and Cell Marker Profiling in High Risk and Relapsed/ Refractory B-Lineage Acute Lymphoblastic Leukaemia
Brief Title: ALaCART-B: Acute Leukemia and Chimeric Antigen Receptor-T Cell Therapy for B-lymphoblastic Leukemia.
Acronym: ALaCART
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/00865
Record Dates: First submitted 2021-05-26; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-04

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood; Lymphoblastic Leukemia; Lymphoblastic Leukemia, Acute Adult; Lymphoblastic Leukemia in Children; CAR; CAR T-Cell-Related Encephalopathy Syndrome
Keywords: B-ALL; CAR-T cell therapy; CAR T-cell therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single arm Phase I Clinical Trial
  Interventions: Biological: CAR T-cell therapy

INTERVENTIONS:
Biological: CAR T-cell therapy — This is a single-centre, phase I study to determine the efficacy and safety of CAR T-cell therapy in patients with high-risk B-ALL, refractory or relapsed B-ALL.

SUMMARY:
The objective of this study is to assess the safety and efficacy of a immunophenotype-adapted approach using CAR T-cells in patients with high-risk, refractory or relapsed B-lineage acute lymphoblastic leukemia (B-ALL).

DETAILED DESCRIPTION:
Patients will receive CART-cells with one or more specificities according to the phenotypic profile of the leukemic cells in each individual patient. This will allow targeting the entire leukemia cell population to induce deeper and more durable remissions. Although it would be possible to administer CART-cells targeting all possible antigens to all patients, this indiscriminate approach would increase the CAR T-cell dose and hence, the risk of toxicity in patients that could be effectively treated with a lower, less toxic, CAR T-cell dose. Moreover, the cost of the procedure increases proportionally with the number of CAR T-cells used, limiting our capacity to enrol other patients. Reducing the number of CART-cells below the dose that we set, will inevitably increase the risk of treatment failure, according to the literature and our own experience.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil the Diagnosis/ Disease define as:

  1. Relapsed B-cell acute lymphoblastic leukaemia/ lymphoma as defined by:

     Bone marrow disease = or > 0.01% by MRD as determined by flow cytometry Or CNS disease as defined as > 5 WBCs in CSF by morphology, or flow cytometric or molecular evidence of blasts or biopsy proven recurrence in the eye or brain.

     Or Extramedullary relapse as defined by morphological evidence of blasts in the testis or any other extramedullary sites
  2. Induction failure as defined by Day 33/ End of induction:

     MRD ≥ 1% by flow cytometry on the Ma-Spore ALL 2020 protocol Or Failure to achieve morphological remission defined as > 5% blasts after standard induction chemotherapy
  3. Refractory disease as defined by:

     MRD ≥ 0.01% by flow cytometry or molecular methods during 2 or more timepoints after induction therapy
  4. Any high risk features including :

     BCR-ABL1, BCR-ABL1-like, - ABL1-r, PDGFRB-r, TCF3-HLF, MLL-r, hypodiploid ALL (< 45 chromosomes), p53 pathogenic mutation as defined by RNA Seq or other molecular methods.
  5. Patients who are unable to tolerate standard chemotherapy due to significant toxicity as well as other comorbidities
* Minimum level of pulmonary reserve defined as grade ≤ 1 dyspnoea and oxygen saturation of > 95% on room air
* Left ventricular systolic function ≥ 28% confirmed by echocardiogram, or left ventricular ejection fraction ≥ 45% confirmed by echocardiogram within 3 months of screening
* Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) performance status ≥ 50 at screening
* Normal Age-adjusted eGFR Creatinine Clearance within 3 months of screening
* Alanine aminotransferase ≤ 5 times the upper limit of normal for age
* Patients with > 99.9% of CD19 expression on blast cells will be eligible for anti-CD19 CAR T-cell infusion.
* Patients with partial or absent CD19 expression (< 99.9%) on blast cells will be eligible to receive combinations of other CAR T-cells depending on the pattern of antigen expression.

Exclusion Criteria:

* Failure to meet any of the inclusion criteria.
* Patients who test positive on urine pregnancy testing and are pregnant or are lactating
* Concomitant genetic syndromes associated with BM failure states, such as Fanconi anaemia, Kostmann syndrome, Schwachman syndrome, or any other BM failure syndrome with the exception of Down syndrome
* Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and no evidence of active disease
* Active or latent hepatitis B or active hepatitis C within 8 weeks of screening, or any uncontrolled infection at screening
* Positive HIV test within 8 weeks of screening
* Grade 2 to 4 acute graft-vs-host disease (GVHD) or extensive chronic GVHD
* Received an investigational medicinal product within 30 days of screening
* Persistent disease or relapse after other forms of CAR-T cell therapy.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participant who are flow cytometry minimal residual disease (MRD) negative at the end of 1 month after CAR T-cell infusion. | 30 days
  MRD levels will be determined by flow cytometry, The target sensitivity of flow MRD is <0.01% when available.

SECONDARY OUTCOMES:
Proportion of participant who are minimal residual disease (MRD) negative with molecular base assay at the end of 1 month after CAR T-cell infusion. | 30 days
  MRD levels will be determined by molecular based MRD. PCR and oncogene fusion transcript (OFT).
Proportion of patient who shows CAR T-cell persistence and presence of B-cell aplasia by immunophenotyping using flow cytometry in bone marrow, peripheral blood and CSF samples at multiple study time points following CAR T cell infusion | 1 month to 5 years
  Flow cytometry will be performed on bone marrow, peripheral blood and CSF samples at multiple study time points following CAR T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Allen Yeoh, M.D, Principal Investigator — National University Hospital, Singapore; Dario Campana, M.D, PhD, Study Director — National University of Singapore
Locations (1):
- Allen Yeoh Eng Juh, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No